CLINICAL TRIAL: NCT01195649
Title: Advanced Renal Cell Carcinoma, With Failure or Unsuitable on Prior Interferon-alpha or Interleukin-2 Based Therapy
Status: Terminated | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15242; NX1010TW (Other: company internal)
Record Dates: First submitted 2010-08-12; First posted 2010-09-06 (Estimated); Last update posted 2019-06-04 (Actual); Status verified 2019-06

CONDITIONS: Carcinoma, Renal Cell
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Patients under daily life treatment according to local drug information

SUMMARY:
The primary objective of this prospective, observational, post-marketing study is to evaluate the patient characteristics, pre-treatment and treatment duration in Renal Cell Carcinoma (RCC) patients who are candidates for systematic therapy and in whom a decision to treat with Nexavar® has been made under real-life practice settings and approved reimbursement restriction in Taiwan. Therefore, the main objective of the study is to collect data on:

Prescription pattern: to determine the factors affecting compliance and duration of treatment with special attention given to education status, demography, disease details, pre-treatment, concomitant medication and other baseline data

Nexavar® treatment and efficacy data

Adverse events using Common Terminology Criteria for Adverse Events (CTCAE) version 4.0

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of advanced Renal Cell Carcinoma (RCC) and decision taken by the investigator to prescribe Nexavar® under Taiwan reimbursement guideline
* Patients must have a life expectancy of at least 8 weeks

Exclusion Criteria:

* Exclusion criteria must follow the approved local product information.
* Patients were lost to follow-up if no follow-up visit and no final assessment of Nexavar® was documented.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Taiwanese patients
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2010-12-13 (Actual); Primary Completion 2012-06-08 (Actual); Study Completion 2012-08-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of Safety and Efficacy of treatments and average doses that are used for patients with Renal Cell Carcinoma (collection of number of adverse events) | After one year
Evaluation of Safety and Efficacy of treatments and average doses that are used for patients with Renal Cell Carcinoma (collection of changes in tumor status) | After one year

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer